CLINICAL TRIAL: NCT01409993
Title: Renin-Angiotensin and Fibrinolysis in Humans: Effect of Long-Term PDE5 Inhibition on Glucose Homeostasis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Aim 1 was stopped by DSMB. Aim 2 was stopped due to ending of funding.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Nancy J. Brown, Hugh J. Morgan Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 110206
Record Dates: First submitted 2011-07-11; First posted 2011-08-04 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Impaired Glucose Tolerance
Keywords: BMI greater than 25; Elevated fasting blood sugar (100-125mg/dL)
MeSH Terms: conditions — Glucose Intolerance | interventions — Sildenafil Citrate; Glucose Clamp Technique

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- sildenafil Aim 1 (Experimental): sildenafil 25 mg p.o. tid
  Interventions: Drug: Sildenafil; Diagnostic Test: Hyperglycemic clamp
- placebo Aim 1 (Placebo Comparator): matching placebo p.o. tid
  Interventions: Drug: Placebo; Diagnostic Test: Hyperglycemic clamp
- sildenafil Aim 2 (Experimental): sildenafil 25 mg p.o. tid
  Interventions: Drug: Sildenafil; Diagnostic Test: Euglycemic clamp
- placebo Aim 2 (Placebo Comparator): matching placebo p.o. tid
  Interventions: Drug: Placebo; Diagnostic Test: Euglycemic clamp

INTERVENTIONS:
Drug: Sildenafil — Sildenafil 25 mg by mouth three times a day for three months
  Arms: sildenafil Aim 1; sildenafil Aim 2
Drug: Placebo — Matching placebo three times a day for three months
  Arms: placebo Aim 1; placebo Aim 2
Diagnostic Test: Hyperglycemic clamp — Subjects with prediabetes will have a baseline hyperglycemic clamp (Aim 1) and then receive sildenafil or placebo for 3 months. Another hyperglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
  Arms: placebo Aim 1; sildenafil Aim 1
Diagnostic Test: Euglycemic clamp — Subjects with prediabetes will have a baseline euglycemic clamp (Aim 2) and then receive sildenafil or placebo for 3 months. Another euglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
  Arms: placebo Aim 2; sildenafil Aim 2

SUMMARY:
The purpose of this study is to determine the effect of chronic PDE5 inhibitor therapy on glucose metabolism in persons with prediabetes.

ELIGIBILITY:
Inclusion criteria:

Age > 18 years and BMI > 25 kg/M2 (> 23 kg/M2 among Asian Americans) Elevated fasting plasma glucose (100-125 mg/dL) IGT (2 hour plasma glucose 140-199 mg/dL) OR metabolic syndrome and/or hemoglobin A1c 5.7-6.4%

Exclusion criteria:

* Diabetes type 1 or type 2, as defined by a fasting glucose of 126 mg/dL or greater, a two hour plasma glucose of 200 mg/dL or greater, or the use of anti-diabetic medication.
* The use of nitrates or any disease that might require the use of nitrates.
* The use of any potent CYP3A4 inhibitor.
* subjects who have participated in a weight-reduction program during the last 6 month or whose weight has increased or decreased more than 2 kg over the preceding 6 months.
* Pregnancy. Women of child-bearing potential will be required to have undergone tubal ligation or to be using barrier methods of birth control.
* Breast-feeding.
* Cardiovascular disease such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy.
* Treatment with anticoagulants.
* Treatment with metformin.
* History of serious neurologic disease such as cerebral hemorrhage, stroke, or transient ischemic attack.
* History or presence of immunological or hematological disorders.
* Diagnosis of asthma.
* Clinically significant gastrointestinal impairment that could interfere with drug absorption.
* Impaired hepatic function (aspartate amino transaminase [AST] and/or alanine amino.

transaminase [ALT] >1.5 x upper limit of normal range)

* Impaired renal function (serum creatinine >1.5 mg/dl).
* Hematocrit <35%.
* Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult.
* Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in

  1 month).
* Treatment with lithium salts.
* History of alcohol or drug abuse.
* Treatment with any investigational drug in the 1 month preceding the study.
* Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study.
* Inability to comply with the protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Ramirez CE, Nian H, Yu C, Gamboa JL, Luther JM, Brown NJ, Shibao CA. Treatment with Sildenafil Improves Insulin Sensitivity in Prediabetes: A Randomized, Controlled Trial. J Clin Endocrinol Metab. 2015 Dec;100(12):4533-40. doi: 10.1210/jc.2015-3415. Epub 2015 Nov 18. PMID 26580240
- [Derived] Ramirez CE, Shuey MM, Milne GL, Gilbert K, Hui N, Yu C, Luther JM, Brown NJ. Arg287Gln variant of EPHX2 and epoxyeicosatrienoic acids are associated with insulin sensitivity in humans. Prostaglandins Other Lipid Mediat. 2014 Oct;113-115:38-44. doi: 10.1016/j.prostaglandins.2014.08.001. Epub 2014 Aug 28. PMID 25173047

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil Aim 1: sildenafil 25 mg p.o. tid
  Administration of Sildenafil: Subjects with prediabetes will have a baseline hyperglycemic (Aim 1) and then receive sildenafil for 3 months. Another hyperglycemic will be performed followed by another 3 months off drug and an oral glucose tolerance test.
- Placebo Aim 1: matching placebo p.o. tid
  Administration of Placebo: Subjects with prediabetes will have a baseline hyperglycemic (Aim 1) and then receive placebo for 3 months. Another hyperglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
- Sildenafil Aim 2: Administration of Sildenafil: Subjects with prediabetes will have a baseline hyperinsulinemic euglycemic (Aim 2) and then receive sildenafil for 3 months. Another euglycemic will be performed followed by another 3 months off drug and an oral glucose tolerance test.
- Placebo Aim 2: Administration of Placebo: Subjects with prediabetes will have a baseline hyperinsulinemic euglycemic (Aim 2) and then receive placebo for 3 months. Another euglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
Period: Overall Study
Arm/Group | Sildenafil Aim 1 | Placebo Aim 1 | Sildenafil Aim 2 | Placebo Aim 2
Started | 25 | 26 | 14 | 13
Completed | 21 | 21 | 11 | 8
Not Completed | 4 | 5 | 3 | 5
Not completed — Adverse Event | 4 | 4 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sildenafil: sildenafil 25 mg p.o. tid
  Administration of sildenafil: Subjects with prediabetes will have a baseline hyperglycemic (Aim 1) or a euglycemic (Aim 2) clamp and then receive sildenafil for 3 months. Another hyperglycemic or euglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
- Placebo: matching placebo p.o. tid
  Administration of placebo: Subjects with prediabetes will have a baseline hyperglycemic (Aim 1) or a euglycemic (Aim 2) clamp and then receive sildenafil or placebo for 3 months. Another hyperglycemic or euglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (10.6) | 51.0 (10.6) | 49.58 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 15 | 13 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 29 | 32 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Insulin Secretion
Description: in the group of subjects undergoing hyperglycemic clamp (Aim 1)
Time Frame: 2.5 hours after 3 months of therapy
Population: Glucose-stimulated insulin secretion from 90 to 120 minutes of hyperglycemic clamp
Measure: Mean (Standard Error); unit: microU/mL
Groups:
- Sildenafil Aim 1: sildenafil 25 mg p.o. tid
  Administration of Sildenafil: Subjects with prediabetes will have a baseline hyperglycemic clamp (Aim 1) and then receive sildenafil for 3 months. Another hyperglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
- Placebo Aim 1: matching placebo p.o. tid
  Administration of Placebo: Subjects with prediabetes will have a baseline hyperglycemic clamp (Aim 1) and then receive placebo for 3 months. Another hyperglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
Arm/Group | Sildenafil Aim 1 | Placebo Aim 1
Number analyzed (Participants) | 21 | 21
microU/mL | 109.4 (85) | 103.1 (67.7)

2. Primary Outcome: Index of Tissue Sensitivity to Insulin
Description: in the group of subjects undergoing hyperglycemic clamp (Aim 1), calculated by dividing the average glucose infusion rate during the last hour of the clamp by the average plasma insulin concentration during the same interval
Time Frame: 2.5 hours after 3 months of therapy
Measure: Mean (Standard Error); unit: (mg/kg/min per microU/mL)*100
Arm/Group | Sildenafil Aim 1 | Placebo Aim 1
Number analyzed (Participants) | 21 | 21
(mg/kg/min per microU/mL)*100 | 6.45 (0.661) | 4.66 (0.661)

3. Primary Outcome: Glucose Infusion Rate
Description: In the group of subjects undergoing euglycemic clamp (Aim 2)
Time Frame: 2.5 hours after 3 months of therapy
Population: one subject in the sildenafil Aim 2 arm has incomplete data from the three-month clamp due to infusion dysfunction
Measure: Mean (Standard Deviation); unit: mL/hr
Groups:
- Sildenafil Aim 2: sildenafil 25 mg p.o. tid
  Administration of Sildenafil : Subjects with prediabetes will have a baseline euglycemic clamp (Aim 2) and then receive sildenafil for 3 months. Another euglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
- Placebo Aim 2: matching placebo p.o. tid
  Administration of Placebo: Subjects with prediabetes will have a baseline euglycemic clamp (Aim 2) and then receive placebo for 3 months. Another euglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
Arm/Group | Sildenafil Aim 2 | Placebo Aim 2
Number analyzed (Participants) | 11 | 7
mL/hr | 140.45 (38.38) | 162.61 (64.49)

4. Secondary Outcome: Fasting Plasma Glucose
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Sildenafil Aim 1: sildenafil 25 mg p.o. tid
  Administration of Sildenafil : Subjects with prediabetes will have a baseline hyperglycemic (Aim 1) and then receive sildenafil for 3 months. Another hyperglycemic or euglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
- Placebo Aim 1: matching placebo p.o. tid
  Administration of Placebo: Subjects with prediabetes will have a baseline hyperglycemic (Aim 1) and then receive sildenafil or placebo for 3 months. Another hyperglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
- Sildenafil Aim 2: sildenafil 25 mg p.o. tid
  Sildenafil: Subjects with prediabetes will have a baseline euglycemic clamp (Aim 2) and then receive sildenafil for 3 months. Another euglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
- Placebo Aim 2: matching placebo p.o. tid
  Placebo: Subjects with prediabetes will have a baseline euglycemic clamp (Aim 2) and then receive placebo for 3 months. Another euglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
Arm/Group | Sildenafil Aim 1 | Placebo Aim 1 | Sildenafil Aim 2 | Placebo Aim 2
Number analyzed (Participants) | 21 | 21 | 11 | 8
mg/dL | 98.6 (11.7) | 96.9 (7.6) | 98.8 (6.5) | 97.5 (11.1)

5. Secondary Outcome: Blood Pressure
Description: Systolic blood pressure
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Sildenafil Aim 1: sildenafil 25 mg p.o. tid
  Sildenafil: Subjects with prediabetes will have a baseline hyperglycemic clamp (Aim 1) and then receive sildenafil for 3 months. Another hyperglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
- Placebo Aim 1: matching placebo p.o. tid
  Placebo: Subjects with prediabetes will have a baseline hyperglycemic clamp (Aim 1) and then receive placebo for 3 months. Another hyperglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
Arm/Group | Sildenafil Aim 1 | Placebo Aim 1 | Sildenafil Aim 2 | Placebo Aim 2
Number analyzed (Participants) | 21 | 21 | 11 | 8
mmHg | 122 (17.2) | 123.1 (14.6) | 114.3 (11.6) | 112.5 (22.6)

ADVERSE EVENTS:
Groups:
- Sildenafil - Aims 1 and 2: sildenafil 25 mg p.o. tid
  Administration of Sildenafil: Subjects with prediabetes will have a baseline hyperglycemic (Aim 1) or a euglycemic (Aim 2) and then receive sildenafil for 3 months. Another hyperglycemic or euglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
- Placebo - Aims 1 and 2: matching placebo p.o. tid
  Administration of Placebo: Subjects with prediabetes will have a baseline hyperglycemic (Aim 1) or a euglycemic (Aim 2) and then receive placebo for 3 months. Another hyperglycemic or euglycemic clamp will be performed followed by another 3 months off drug and an oral glucose tolerance test.
Arm/Group | Sildenafil - Aims 1 and 2 | Placebo - Aims 1 and 2
Serious Adverse Events (participants affected / at risk) | 1/39 | 0/39
Other Adverse Events (participants affected / at risk) | 32/39 | 25/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil - Aims 1 and 2 (N=39) | Placebo - Aims 1 and 2 (N=39)
hypertension and bradycardia (Cardiac disorders) | 1 (38) | 0 (0) — Patient hospitalized with systolic blood pressure of 190 mm Hg and bradycardia. During hospitalization tested positive for a sympathomimetic drug. Subject was withdrawn from study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil - Aims 1 and 2 (N=39) | Placebo - Aims 1 and 2 (N=39)
headache (Nervous system disorders) | 15 | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 10
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Gastrointestinal symptoms (Gastrointestinal disorders) | 11 | 6
Flushing (Vascular disorders) | 5 | 1
Lightheadeness (General disorders) | 4 | 1
Edema (General disorders) | 2 | 0
Weight gain (General disorders) | 2 | 0
Smell or taste abnormality (Nervous system disorders) | 2 | 0
abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 2
transient numbness (Surgical and medical procedures) | 0 | 2 — numbness related to IV placement e.g.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes